CLINICAL TRIAL: NCT05205889
Title: A Mobile Intervention on Values in Chronic Pain Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Jenny Riecke, Principal Investigator Jenny Riecke, Philipps University Marburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCA0222
Record Dates: First submitted 2021-12-21; First posted 2022-01-25 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Chronic Pain Syndrome

STUDY DESIGN:
Intervention Model Description: Single case analysis with 10-17 pre-measurement time points; 10 measurement time points during the intervention; and one post-measurement.
Masking Description: No masking is required, as participants are fully informed about the purpose of the study. Since there is only one arm, masking of the investigators is also not necessary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile based values intervention for people with chronic pain (Experimental)
  Interventions: Behavioral: Mobile intervention on values and goals in patients with chronic pain.

INTERVENTIONS:
Behavioral: Mobile intervention on values and goals in patients with chronic pain. — The protocol consists of 10 daily sessions, 10-20 Minutes each. After each session participants will complete daily measures. Participants will learn about values and a values based life. Further they will identify their own values and are encouraged to set a goal to pursue those values. Based on this, barriers to achieving goals are explained and a corresponding commitment will be made.

SUMMARY:
The study aims to test a mobile intervention on values and goals in chronic pain patients. The cognitive behavioral intervention is a 10-day course in which participants complete a brief intervention each day (about 10-20 minutes a day). The content of the intervention includes the definition of values; development of individualized values and personal value-oriented goals; and implementation of personal goals in every day life. To assess the effectiveness of the intervention, we use a multiple baseline single case design. Baseline measurements will be assessed daily between 10 and 17 days (the exact number will be randomized). Daily measurements will continue during the intervention. After the intervention, another post measurement will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Chronic, non-tumor related back pain (pain for at least 6 months)
* Ownership of a smartphone
* Numeric Rating Scale for pain result of ≥ 4

Exclusion Criteria:

* High cognitive impairment (e.g., intellectual disability)
* Currently in psychotherapeutic treatment
* Initiation of pain-focused treatment during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Subjects can self-assign their gender.
Enrollment: 30 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Pain intensity | Pain intensity is assessed daily from baseline to the end of treatment (resulting in 20-27 measuring time points)
  Numerical Pain Rating Scale (NPRS) Minimum value: 0; Maximum value: 10 (higher scores indicate higher pain intensity)

SECONDARY OUTCOMES:
Change in psychological well-being | Psychological well-being is assessed daily from baseline to the end of treatment (resulting in 20-27 measuring time points)
  The five-item WHO Well-Being Index (WHO-5) Minimum value: 0; Maximum value 10 (range is adapted for the study; higher scores indicate higher psychological well-being)
Change in chronic pain acceptance | Chronic Pain Acceptance is assessed daily from baseline to the end of the study (resulting in 20-27 measuring time points)
  Chronic Pain Acceptance Questionnaire (CPAQ) Minimum value: 0; Maximum value: 10 (range is adapted for the study; higher scores indicate higher pain acceptance)
Change in engaged living | Engaged Living is assessed daily from baseline to the end of the study (resulting in 20-27 measuring time points)
  Engaged Living Scale (ELS) Minimum value: 0; Maximum value: 10 (range is adapted for the study; higher scores indicate higher engaged living)
Change in pain catastrophizing | Pain Catastrophizing is assessed daily from baseline to the end of the study (resulting in 20-27 measuring time points)
  Pain Catastrophizing Scale (PCS) Minimum value: 0; Maximum value: 10 (range is adapted for the study; higher scores indicate higher catastrophizing)
Change in psychological flexibility | Psychological Flexibility is assessed daily from baseline to the end of the study (resulting in 20-27 measuring time points)
  Acceptance and Action Questionnaire 2 (AAQ-2) Minimum value: 0; Maximum value: 10 (range is adapted for the study; higher scores indicate lower psychological flexibility)
Change in self-efficacy | Self-efficacy is assessed daily from baseline to the end of the study (resulting in 20-27 measuring time points)
  Pain Self-efficacy Questionnaire (PSEQ) Minimum value: 0; Maximum value: 10 (range is adapted for the study; higher scores indicate higher self-efficacy)

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, PhD, Principal Investigator — Philipps University Marburg
Locations (1):
- University of Marburg, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared upon request.